CLINICAL TRIAL: NCT02042469
Title: Awareness and Attitude of Cancer Patients About Participation in Clinical Research (CR) in Saudi Arabia
Status: Completed | Type: Observational
Sponsor: National Guard Health Affairs (Other Government)
Responsible Party: Sponsor
Other Study IDs: Awareness
Record Dates: First submitted 2014-01-15; First posted 2014-01-22 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Oncology [See Also, Affected System]
Keywords: awareness, clinical research, Saudi arabia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Survey: Cross-sectional survey will be carried out using an interview questionnaire composed of close-ended questions to be completed by trained research coordinator.

SUMMARY:
Enrollment of patients in CR may be impacted by their levels of awareness and attitude toward participation. Our study aims at assessing the awareness and willingness to participate in CR and identifying the barriers and influencing factors for participation.

A cross-sectional study was performed using an interview-based questionnaire composed of close-ended questions conducted by trained research coordinators. Descriptive statistics, univariate and multivariate analyses were applied.

DETAILED DESCRIPTION:
Clinical Trials are essential for the identification of effective therapies in modern medicine. As the biomedical understanding of diseases increases, a growing number of new opportunities will require increasing numbers of patients agreeing to participate in a clinical trial

Public awareness about the need for clinical research and the benefit beyond participation is important. Although the main objective of clinical trials is to provide a high standard of care and help in advancement of medical knowledge, only a small portion of patients receive treatment as part of a formal clinical trial

Misconceptions about clinical trials are frequent, primarily due to lack of adequate information from the treating physician; the complexity of the study procedure; preferences of patients regarding a particular treatment or no treatment; uncertainty and the experimental nature of a clinical trial (additional side effects, less known about the treatment) and concern about confidential information are some of the significant barriers to participation. Healthy individuals and patients do not have the same perception, since patients have stressed and vulnerable feelings after diagnosis of their illness having a negative impact on patient's attitude towards a trial.

The ability to recruit patients for future clinical trials will depend, in part, on understanding the barriers of participation in clinical trials. Unfortunately, there is no data about the public awareness and attitudes toward participation in clinical trials in Kingdom of Saudi Arabia. It is the purpose of this study to address this issue to create some baseline data to increase the accrual rate of clinical trials.

ELIGIBILITY:
Inclusion Criteria:

Adult patient (18 years and above) with cancer diagnosis. Adult patients who are treated services at King Abdulaziz Medical City (KAMC), National Guard Health Affairs(NGHA) Riyadh Willing to complete the survey questionnaire

Exclusion Criteria:

Patients who refuse to complete the survey questionnaire

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study is planned to take place among Oncology patients ( inpatient and outpatient).
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2011-04; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Measure the awareness and attitudes | 2 years
  To study the Awareness and Attitudes of Saudi adult cancer patients towards participation in clinical research.

SECONDARY OUTCOMES:
assess knowledge | 2 years
  To assess the knowledge of cancer patients about the clinical research process. To assess cancer patients willingness to participate in clinical research. To identify the patients barriers to clinical research participation.

CONTACTS AND LOCATIONS:
Overall Officials: Nagham RZ Sheblaq, CCRP, Principal Investigator — King Abdul Aziz Medical City for National Guard
Locations (1):
- King Abdul Aziz Medical City for National Guard, Riyadh, Saudi Arabia